CLINICAL TRIAL: NCT03271944
Title: Fractional Handpiece With CO2 Laser: Fractional Ablative Laser Treatment of Vulvovaginal Atrophy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SHERRY Thomas (Other)
Collaborators: Perigree Medical (Unknown)
Responsible Party: Sponsor-Investigator, SHERRY Thomas, Principal Investigator, The American Association of Female Pelvic Medicine Specialists, Inc.
Organization: The American Association of Female Pelvic Medicine Specialists, Inc. (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20161370
Record Dates: First submitted 2017-08-29; First posted 2017-09-05 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Vulvovaginal Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Single group 30 post menopause females. (Other)
  Interventions: Device: CO2 Laser Treatment

INTERVENTIONS:
Device: CO2 Laser Treatment — Fractional handpiece with CO2 laser: Fractional Ablative laser Treatment of Vulvovaginal Atrophy

SUMMARY:
To assess the feasibility and efficacy of the CO2 fractional handpiece in the treatment of vulvovaginal atrophy (VVA) in post-menopausal women and its effect on the patient VHIS(vaginal health index core). The primary endpoint is to assess the change in the vaginal dryness by means of a visual analogic scale (10 cm VAS).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the use of a CO2 laser (EdgeTM CO2 Laser) with a fractional handpiece made specifically for the vagina to possibly restore the normal physiological conditions of the vagina, thus reducing the symptoms of VVA. The EdgeTM CO2 Laser and general fractional handpiece is approved by the FDA for ablative skin resurfacing (for example, treating fine lines and wrinkles, acne and surgical scars, skin pigmentation and discoloration, sun damage, pre-cancerous as well as benign lesions and uneven skin texture). The fractional handpiece used in this study for the treatment of VVA is experimental and has not been approved by the FDA for vaginal dryness associated with menopause.

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting the following inclusion criteria may participate:

  * Healthy non-smoking post menopausal women with absence of menstruation of at least 12 months
  * Exhibiting VVA symptoms
  * Prolapse staged < II, according to the pelvic organ prolapse quantification (ICS-POP- Q) system
  * Have not had procedures in the anatomical area through 6 months prior to treatment
  * Understand and accept the obligation and is logistically able to present for all scheduled follow-up visits

Exclusion Criteria:

* Subjects meeting any of the following criteria will be excluded from participation:

  * Acute or recurrent urinary tract infection (UTI), or genital infection (e.g. herpes candida).
  * Prolapse staged ≥ II, according to the pelvic organ prolapse quantification (ICS-POP- Q) system
  * Any serious disease, or chronic condition, that could interfere with the study compliance
  * Previously undergone reconstructive pelvic surgery
  * Have used vaginal creams, moisturizers, lubricants or homeopathic preparations for at least 3 months
  * A history of thrombophlebitis
  * A history of acute infections
  * A history of heart failure
  * Received or is anticipated to receive antiplatelets, anticoagulants, thrombolytics, vitamin E or anti inflammatories within 2 weeks pre treatment
  * Any medical condition, that, in the investigator's opinion would interfere with the patient's participation in the study
  * Taking medications that are photosensitive
  * A history of keloid formation

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-12-29 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Fractional handpiece with CO2 laser: Fractional Ablative laser Treatment of Vulvovaginal Atrophy (VVA). | 9 month
  The purpose of this study is to evaluate efficacy and safety of CO2 laser (EdgeTM CO2 Laser) with a fractional headpiece in the treatment of vulvovaginal atrophy (VVA) in post- menopausal women and its effect on the patient VHIS (vaginal health index score). The primary endpoint is to assess the changes in the vaginal dryness by mean of a visual analog scale (10 cm VAS).

CONTACTS AND LOCATIONS:
Locations (1):
- The American Association of Female Pelvic Medicine Specialists, Inc., Agoura Hills, California, United States

IPD SHARING:
Plan to Share IPD: Undecided